CLINICAL TRIAL: NCT06570005
Title: Evaluating a Water Quality Assurance Fund Intervention in Ghana and Kenya
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Aquaya Institute (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Conrad N. Hilton Foundation (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other); Kwame Nkrumah University of Science and Technology (KNUST) (Unknown); Water Mission (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: REAL-Water Assurance Fund
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Water Quality; Water Treatment; Knowledge; Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Stepped-wedge Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Assurance Fund Intervention Arm 1 (Experimental): In this study arm, intervention activities will start after initial baseline data collection.
  Interventions: Other: Water Quality Assurance Fund
- Assurance Fund Intervention Arm 2 (Experimental): The intervention activities are the same as those described in Arm 1. However, in this study arm, the intervention activities will start 6 months later than those in Arm 1. This arm will serve as a controlled comparison during those initial 6 months.
  Interventions: Other: Water Quality Assurance Fund
- Assurance Fund Intervention Arm 3 (Experimental): The intervention activities are the same as those described in Arm 1. However, in this study arm, the intervention activities will start 12 months later than those in Arm 1. This arm will serve as a controlled comparison during those initial 12 months.
  Interventions: Other: Water Quality Assurance Fund
- Non-randomized Arm (Experimental): In Ghana only, there is a fourth study arm that will receive the intervention one month prior to Arm 1. This group was non-randomly selected and will primarily serve to support qualitative lessons learned from the Assurance Fund program.
  Interventions: Other: Water Quality Assurance Fund

INTERVENTIONS:
Other: Water Quality Assurance Fund — * At the water system level: Written legal agreements between water systems, centralized laboratories, and the organization facilitating the Assurance Fund will provide water systems with regular water quality testing and provide laboratories a guarantee of payments if water systems fail to pay for testing services on time (for up to three concurrent unpaid invoices). Regular debrief meetings will be held with water operators and local government authorities to discuss test results and water treatment options, and to encourage water systems to share water quality information with their consumers. Technical guidance to improve water treatment will be provided, if requested by water system operators or local government authorities.
  * At the community level: Community engagement, primarily at the onset, to inform the community about the water quality testing program and answer questions.

SUMMARY:
The objective of this study is to evaluate the effects of a novel financial and capacity strengthening intervention (the 'Water Quality Assurance Fund' program) on water safety management in rural Ghana and Kenya. The investigators hypothesize the intervention will improve water system operator knowledge, chlorination practices, and water quality at the point of collection, as well as improve consumer satisfaction, awareness, and willingness-to-pay for water that is tested and treated.

DETAILED DESCRIPTION:
Regular water quality monitoring by water suppliers is essential for maintaining adequate treatment processes and verifying safe water quality to protect public health. Yet, many small water suppliers are unable to conduct regular water quality tests due to financial, logistical, and capacity constraints. The goals of the Water Quality Assurance Fund program are to address these constraints by incentivizing established laboratories to extend their services to these smaller water systems and, in parallel, promote the use of water quality data for better water safety management.

The objective of this study is to evaluate the effects of a novel financial and capacity strengthening intervention (the 'Water Quality Assurance Fund' program) on water safety management in rural Ghana and Kenya. As part of the intervention, written legal agreements between water systems, centralized laboratories, and the organization facilitating the Assurance Fund will provide water systems with regular water quality testing and provide laboratories a guarantee of payments if water systems fail to pay for testing services on time. The Assurance Fund program will also deliver capacity strengthening, technical guidance, and community sensitization activities.

The investigators hypothesize the intervention will improve water system operator knowledge, chlorination practices, and water quality at the point of collection, as well as improve consumer satisfaction, awareness, and willingness-to-pay for water that is tested and treated. A secondary aim is to assess implementation challenges and enabling factors associated with the expansion of water testing services by existing professional water quality laboratories to rural water suppliers.

ELIGIBILITY:
Eligibility to receive the intervention was determined by water system criteria:

Inclusion Criteria:

* The district or county government was interested in participating in the Assurance Fund program and water systems within the district/county were accessible to a partner central laboratory that was able to provide water sample collection and testing services for a fee.
* Water systems were functional.
* Water systems were piped water systems (Kenya, Ghana) or mechanized boreholes with a single tapstand (Ghana).
* Water systems could afford regular water quality testing from the selected laboratory.

Exclusion Criteria:

* Water systems did not meet above inclusion criteria.

To be eligible to participate in household surveys, participants need to be at least 18 years of age and a customer of a eligible water system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Adequate free chlorine residual in water at the point of collection | Baseline, 6-months, 12-months, 18-months, 24-months
  Free chlorine residual in water at the point of collection above targeted levels of 0.2 mg/L.

SECONDARY OUTCOMES:
Detectable free chlorine residual in water at the point of collection | Baseline, 6-months, 12-months, 18-months, 24-months
  Free chlorine residual in water at the point of collection above detectable levels of 0.1 mg/L.
E. coli in water at the point of collection | Baseline, 6-months, 12-months, 18-months, 24-months
  E. coli in water at point of collection (binary and categorical).
Water system operator knowledge | Baseline, 12-months, 24-months
  Water system operator knowledge related to water quality (score out of 32 points on a knowledge assessment).
Consumer awareness | Baseline, 12-months, 24-months
  Household respondent is aware enrolled water is tested or treated
Consumer satisfaction | Baseline, 12-months, 24-months
  Household respondent is satisfied with water supplier. They will be considered satisfied if they report they are either very satisfied or somewhat satisfied with the water supplier. They will be considered dissatisfied if they report they are either very dissatisfied or somewhat dissatisfied with the water supplier.
Willingness-to-pay | Baseline, 12-months, 24-months
  Stated willingness-to-pay for treated and tested water for standpipe and private tap users (% increase and absolute increase in local currency).
Adequate free chlorine residual in household stored water | Baseline, 12-months, 24-months
  Free chlorine residual in household stored water above targeted levels of 0.2 mg/L.
Detectable free chlorine residual in household stored water | Baseline, 12-months, 24-months
  Free chlorine residual in household stored water above detectable levels of 0.1 mg/L.
E. coli in household stored water | Baseline, 12-months, 24-months
  E. coli in household stored water (binary and categorical).

OTHER OUTCOMES:
Water system chlorination frequency | Baseline, 6-months, 12-months, 18-months, 24-months
  Water system operator reports weekly chlorinating frequency.
Water system revenue | Baseline, 6-months, 12-months, 18-months, 24-months
  Revenue reported by water systems.
Households use of enrolled water for drinking | Baseline, 12-months, 24-months
  Households use of enrolled water for drinking (binary).

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Bauza, PhD, Principal Investigator — The Aquaya Institute
Locations (2):
- The Aquaya Institute, Accra, Ghana
- The Aquaya Institute, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available.
Supporting Information: Study Protocol, SAP, ICF